CLINICAL TRIAL: NCT01527890
Title: Effect of Intravenous Patient-controlled Analgesia (IV-PCA) With Fentanyl in Adults for Acute Postoperative Pain Control
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Yon Hee Shim, Yonsei University College of Medicine, Yonsei University
Other Study IDs: 3-2011-0238
Record Dates: First submitted 2012-01-27; First posted 2012-02-07 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Nausea; Vomiting
Keywords: intravenous patient-controlled analgesia; IV PCA
MeSH Terms: conditions — Nausea; Vomiting | interventions — Fentanyl

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Drug: Fentanyl — intravenous patient-controlled analgesia

SUMMARY:
In this retrospective study, the investigators examined incidence and risk factors of postoperative nausea and vomiting (PONV) in patients with fentanyl-based intravenous patient-controlled analgesia (IV-PCA).

ELIGIBILITY:
Inclusion Criteria:

1. Adults between 20 to 60 years old
2. Date from 1st, May 2011 to 31st, October 2011
3. Patients with fentanyl based intravenous patient-controlled analgesia for postoperative pain control

Exclusion Criteria:

1. Reoperation within 48 hours
2. Patients who cannot express numerical rating scale for pain due to sedation

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with Intravenous Fentanyl Patient-controlled Analgesia for postoperative pain control
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2012-02; Primary Completion 2012-09 (Estimated); Study Completion 2012-10 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea